CLINICAL TRIAL: NCT01293253
Title: Danish: Integreret Motion på Arbejdspladsen (IRMA) English: Implementation of Exercise at the Workplace
Brief Title: Effect of Daily Stair Walking on Cardiovascular Health
Acronym: IRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Lars L. Andersen, Senior Researcher, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRMA01
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Cardiovascular Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stair walking (Experimental): Participants of this group is encouraged to use the stairs for 10 minutes a day at the workplace
  Interventions: Behavioral: Stair walking
- Control (Active Comparator): Receives a health examination before and after the intervention period, and are advised to stay active
  Interventions: Behavioral: Stair walking

INTERVENTIONS:
Behavioral: Stair walking — Participants of the stair group is encouraged to use the stairs for 10 minutes a day at the workplace. Participants of the control group receive a health examination before and after the intervention period, and are advised to stay active

SUMMARY:
Many adults find it difficult to perform physical exercise during leisure. The workplace may provide an optimal setting to encourage a healthier lifestyle. This study investigates the effect of daily stair walking at the workplace on cardiovascular health.

The main hypothesis is that daily stair walking for 10 weeks compared with a control group results in increased aerobic fitness.

ELIGIBILITY:
Inclusion Criteria:

* office worker

Exclusion Criteria:

* life threatening disease
* pregnancy

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Aerobic fitness | before and after the 10 week intervention
  Watt-max test on a Monark bicycle ergometer

SECONDARY OUTCOMES:
Blood pressure | before and after the 10 week intervention
Questionnaire-based data | before and after the 10 week intervention
  working conditions, perceived health, tiredness and energy, physical activity
Heart Rate Variability | Before and after the 10 week intervention
  HRV during rest is measured during a standardized test (5 min supine, 5 minute upright, 5 minute supine)

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — National Research Centre for the Working Environment, Denmark
Locations (1):
- Lægemiddelstyrelsen, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen LL, Sundstrup E, Boysen M, Jakobsen MD, Mortensen OS, Persson R. Cardiovascular health effects of internet-based encouragements to do daily workplace stair-walks: randomized controlled trial. J Med Internet Res. 2013 Jun 21;15(6):e127. doi: 10.2196/jmir.2340. PMID 23793032